CLINICAL TRIAL: NCT01136668
Title: Transversus Abdominis Plane Block in Children Undergoing Ostomy Surgery: A Prospective Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane Block in Children Undergoing Ostomy Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit adequate number of subjects
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000014754
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Anesthesia; Ostomy
Keywords: pediatrics; Transversus Abdominis Plane Block; Ostomy Surgery; Anesthesia; Regional Anesthetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Bupivacine-TAP block
  Interventions: Procedure: Transversus Abdominis Plane Block
- Control Group (Active Comparator): Bupivacaine- wound infiltration
  Interventions: Procedure: Standard

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block — A high frequency (5-10 mHz) ultrasound probe (Sonosite Micromaxx, Licence No 12407) will be placed on the flank at the midpoint between the iliac crest and lower costal margin. The three muscle layers of external oblique, internal oblique, and transversus abdominis will be visualized. A 22G short-bevel block needle will be advanced in an anterior-to-posterior direction, in-plane with the probe, until the tip is visualized in the transversus abdominis plane. After negative aspiration, 0.4 ml/kg of bupivacaine 0.25% with 1:200,000 epinephrine will be injected. The total dose of bupivacaine will not exceed 2 mg/kg and the total volume will not be more than 20 ml.
  Arms: Treatment group
Procedure: Standard — Circumferential subcutaneous infiltration of the ostomy wound with bupivacaine 0.25% with 1:200 000 epinephrine 0.4 ml/kg by the surgeon after skin closure.
  Arms: Control Group

SUMMARY:
The primary objective of this study is to determine if the use of Transversus Abdominis Plane (TAP) blocks reduce early postoperative opioid requirements.

DETAILED DESCRIPTION:
Revision or closure of ostomy is a common elective surgical procedure at The Hospital for Sick Children. A retrospective audit conducted at SickKids demonstrated significant intraoperative opioid use and significant requirements for rescue opioids in recovery.

Concerns exist regarding the relative merits of opioid use in abdominal surgery. Opioids may decrease bowel motility leading to the increased incidence and duration of postoperative ileus. They may be associated with increased rates of post-operative nausea and vomiting and pruritus. Lastly children may under-report their pain or pain may not be recognized by medical staff leading to inadequate provision of analgesia. This suggests that the use of a regional technique may benefit children undergoing revision of ostomy.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing revision or closure of ostomy
* American Society of Anesthesiologists Classification 1-3.
* age ≥ 3 months

Exclusion Criteria:

* children undergoing an additional surgical procedure (e.g. circumcision) at an anatomical location not covered by a one-sided/ unilateral TAP block, during the same anesthetic
* children in whom a TAP block is contraindicated, i.e. surgical scar or distorted anatomy at the site of injection
* postoperative admission to the intensive care unit
* children with a known allergy to bupivacaine
* children with a history of chronic abdominal pain
* use of opioid analgesics prior to surgery
* pregnancy
* impaired renal function
* impaired hepatic function
* known impaired cardiac function
* hypersensitivity to sodium metabisulfite

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 2 (2) | 7 (11) | 5 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Morphine Requirement
Description: The primary endpoint will be the proportion of children in each group requiring two or more (≥ 2) boluses of morphine in the PACU.
Time Frame: within the first 48 hours after surgery
Population: Data not collected
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No